CLINICAL TRIAL: NCT01839045
Title: Breast Cancer Biomarker Sample Collection for the DtectDx Assay Proof of Concept
Brief Title: Breast Cancer Biomarker Sample Collection for the dtectDx Assay Verification
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Provista Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: dtectDx-Breast-001; ProvistaDx (Other: ProvistaDx)
Record Dates: First submitted 2013-04-05; First posted 2013-04-24 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: Woman; Breast Cancer; Cancer; Mammogram; Ultrasound; Imaging; Biomarkers; ACR BI RAD Category 3; ACR BI RAD Category 4
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — At each visit, 35mL or 2 1/2 tablespoons of blood will be drawn from your arm.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Breast Cancer: ACR BI-RAD Category 3 or 4 result

SUMMARY:
The major purpose of this study is to evaluate a laboratory developed test that measures multiple breast cancer-specific biomarker proteins in your blood samples. The biomarker results along with your personal medical profile will be evaluated to determine your risk for the presence of a malignancy in the breast as compared to your breast evaluation assessment conducted by your physician.

DETAILED DESCRIPTION:
As part of the study, 35 mL or 2 1/2 tablespoons of blood will be drawn from your arm at each study visit.

This study has 2 visits. Visit 1 will take about 1 hour. Visit 2 is a follow up visit at 6 months taking about 1 hour.

Visit 1- Screening and Blood Collection:

The following procedures will be done at the clinical research facility:

* The study doctor and/or study staff will explain the study and all the study procedures.
* You will be asked to review, sign and date this informed consent before any procedures are done.
* The study doctor and/or study staff will ask you questions about your health status and medical history and record this information.
* 35 mL or 2 ½ tablespoons of blood will be collected from your arm.
* The samples will not be labeled with your name but a unique identification code, which means they will be given a number which can be linked to you.

Visit 2 - Follow up:

If you have been diagnosed with cancer between visit 1 and visit 2, you will not be required to complete visit 2. If you have been diagnosed with LCIS or DCIS, you will be requested to return for visit 2. Otherwise you will return to the center for visit 2.

The following procedures will be performed:

* You will have a follow-up breast evaluation performed. Your follow-up breast evaluation may occur prior to Visit 2 if you have it performed at a different facility or it may be performed during this study visit.
* The study doctor and/or study staff will assess your health and medical history.
* 35 mL or 2 1/2 tablespoons of blood will be collected from your arm.
* The samples will not be labeled with your name but a unique identification code, which means they will be given a number which can be linked to you.

Your blood sample will be sent to the study Sponsor, Provista Diagnostics, Inc. for testing.

The test results will not be reported back to the study doctor and will not be used to determine or change your treatment. This testing will be done in addition to any routine testing that your study doctor performs. You will not receive the results of these tests.

Up to 350 subjects will take part in this study. Patients will be enrolled at one of seven sites.

ELIGIBILITY:
Inclusion Criteria:

* Adult women from 25 years of age to below 50 years of age
* Breast evaluation results of ACR BI-RADS® Category 3 or 4 by imaging and physicians clinical and radiological evaluation
* Study visit and blood collection within 3 weeks (21 days) of ACR BI-RADS assessment
* Patient agrees to return for diagnostic follow-up and blood collection at 6 months unless a positive cancer diagnosis is made between study visits 1 and 2. Individuals diagnosed with LCIS and DCIS will agree to return for visit 2
* Samples collected under IRB approval and Informed Consent
* Testing performed under IRB approval or waiver (as applicable)

Exclusion Criteria:

* Adults from 50 years of age or older and below 25 years of age
* Final breast evaluation results other than a ACR BI-RADS Category 3 or 4
* Subjects that have had a breast biopsy performed at any time prior to the study visit
* Samples not collected under IRB approval and Informed Consent
* Testing not performed under IRB approval or waiver (as applicable)
* Prior breast cancer diagnosis.

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary Care Clinics
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Training | Baseline
  Part I: Establish an acceptable algorithm for generation of a single numerical score from the combination of the 5 cancer biomarkers that comprise the dtectDX-Breast Assay Part II: Define a numerical score cutoff that differentiates malignant from nonmalignant breast cancer in this population of woman.
Blinded Validation | 6 months
  Demonstrate proof-of-concept for use of the dtectDx-Breast Assay to assess likelihood of breast cancer malignancy in conjunction with the physicians clinical and radiological evaluations.

SECONDARY OUTCOMES:
Clinical Sensitivity/Specificity | Baseline
  Demonstrate the numerical score, collaborated via proprietary algorithm (greater then 60 is an elevated score, less then 60 is a normal score), for the dtectDx-Breast Assay increases the likelihood of malignant breast cancer detection when used adjunctively with the assessment of BI-RADS Categories 3 and 4 compared to the assessment of BI-RADS Categories 3 and 4 alone.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Banner Health, Phoenix, Arizona
  - Sutter Institute, Sacramento, California
  - Scripps, San Diego, California
  - Sansum Clinic, Santa Barbara, California
  - Lahey Clinic, Peabody, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Rhode Island Hospital, Providence, Rhode Island
  - Avera Research Institute, Sioux Falls, South Dakota

REFERENCES:
- See also: Related Info — http://www.provistadx.com